NCT Number: NCT02536963

**Study Title:** Improving Quality Vision Outcomes in Managed Care Setting While Reducing Cost

by Use of Accurate, Automated Screening

**Document:** Informed Consent

Date Created: August 2015

## I. Informed Consent Form

| KAISER FOUNDATIO | ON HOSPITALS | PATIENT'S | S NAME: |
|---|---|---|---|
| SOUTHERN CALIFO<br>MEDICAL GROUP | RNIA PERMANENTE | | |
| INFORMED CONSENT TO PARTICIPATE IN A RESEARCH STUDY: Improving quality vision outcomes in the managed care setting while reducing cost by use of accurate, automated screening | | | |
| SPONSOR: | National Institutes | of Health (I | NIH) |
| INVESTIGATOR: | | | |
| TELEPHONE: | | | |

Your child is being invited to be in a research study. The purpose of this form is to give you detailed information about this study. Our goal is for you to understand:

- that taking part in a research study is entirely voluntary,
- the reason we are doing the study,
- what will happen to you if you decide to be in the study, and
- what will happen to you if you decide not to be in the study.

You can ask the study staff any questions at any time. You can take this form home to think about the study or talk to family and friends about it.

Participating in a research study is not the same as getting regular medical care. Therefore, it is important that you understand the difference between the regular care you get from your doctor and what is involved in this research study.

The purpose of regular medical care is to improve your child's health. The purpose of a research study is to gather information to advance medicine. There is no guarantee that your child will directly benefit from the research study. Your child's study doctor and the research staff assisting your child's study doctor must follow the requirements of the research study. Being in this study does not replace your child's regular medical care.

Kaiser Permanente is being paid by the study sponsor, National Eye Institute (a branch of the NIH), to conduct this research.

KPSC IRB Board Approved: 08/18/2015

IRB NUMBER: 10764
IRB APPROVAL DATE: 08/18/2015
IRB EXPIRATION DATE: 07/25/2016

## II. Enrollment Form

| Vision Screening Study | | |
|---|---|---|
| Participant Enrollment Form | | |
| Form #1 Version: 12/5/2014 | | |
| SECTION A: GENERAL INFORMATION | | |
| A1. | Study ID number | |
| A2. | A2. Visit Date: MM/DD/YYYY / / | |
| A3. Initials of person completing form: | | |
| A4. Date Form Completed: MM/DD/YYYY/// | | |
| SECTION B: Demographics | | |
| B1. | Name | |
| B2. | KP# | |
| В3. | Date of Birth: | MonthDayYear |
| B4. | Gender: | MaleFemale |
| B5. | Race: | American Indian/Alaska Native |
| | | Asian |
| | Native Hawaiian or Other Pacific Islander | |
| | Black or African American | |
| | | White |
| | | More than one race |
| B6. | Ethnicity: | Hispanic or Latino |
| | | Not Hispanic of Latino |
| B7. | Corrective Ler | ns Use:No |
| B8. | History of Ocu | ılar Disease:YesNo |
| | Specify | if yes: |

## III. Eligibility Form

| SECTION A: GENERAL INFORMATION | | | |
|---|---|---|---|
| A1. Study ID number | | | |
| A2. \ | Visit Date: MM/DD/Y | | |
| A3. I | nitials of person completing form: | | |
| A4. I | Date Form Completed: MM/DD/YYYY/// | | |
| SEC | TION B: ELIGIBILITY CHECKLIST | | |
| | Criteria | Yes | No |
| B1. | Is the subject older or equal to 2 years of age, and less than 6 years of age? | | |
| | If yes, continue to B2. | | |
| | If no, subject is not eligible for study. | | |
| B2. | Does the subject have any apparent developmental delay or cognitive | | |
| | deficit? | | |
| | If yes, subject is not eligible for study. | | |
| | If no, continue to B3. | | |
| В3. | Does the subject have any visually obvious ocular conditions (cosmetically | | |
| | obvious strabismus, ptosis, gross nystagmus, eye infection, etc.) that would | | |
| | warrant specialist referral? | | |
| | (Children wearing glasses are not to be excluded, unless they have the | | |
| | visually obvious conditions listed.) | | |
| | If yes, subject is not eligible for study. | | |
| | If no, subject is eligible for study. | | |
| | Is subject eligible for study? | | |
| L | | <u>.I.</u> | I |
| Name | e of person conducting screening (first & last): | | |
| Signa | ature: | | |
| Date: | | | |